CLINICAL TRIAL: NCT02017665
Title: Singapore Neurologic Infections Program
Acronym: SNIP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: Tan Tock Seng Hospital (Other); Duke-NUS Graduate Medical School (Other); Changi General Hospital (Other); Khoo Teck Puat Hospital (Other); National University Health System, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/374/E
Record Dates: First submitted 2013-11-04; First posted 2013-12-23 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Central Nervous System Infections
Keywords: encephalitis; viral infections; central nervous system
MeSH Terms: conditions — Central Nervous System Infections; Encephalitis; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood, cerebrospinal fluid, throat/nasopharyngeal swabs, urine and rectal swabs or stool samples wil be stored for maximum 10 years.All samples will be de-identified and coded
Oversight: Data Monitoring Committee: No

SUMMARY:
Worldwide, central nervous system infections such as inflammation of brain (encephalitis), inflammation of meninges (meningitis) and sudden onset of weakness of muscles which maybe infectious in origin result in significant illness and death and healthcare costs. Vast majority of central nervous system infections remain without an identifiable cause. There is also concern about new and emerging infections.

This study thus intends to fill in the gaps in knowledge with regards to central nervous system infections in Singapore to give a thorough description of burden of causes of central nervous system infections and detection of outbreaks of new pathogens. Patients suspected of central nervous system infection will be recruited from 5 restructured Singapore hospitals and their blood and other clinical specimens will be sent for testing. Patients will also be followed up to assess long term outcomes and socio-economic costs of these infections. This will help clinicians, policymakers and public health officials in estimating financial and societal costs of CNs infections in Singapore.

DETAILED DESCRIPTION:
The study aims to:

1. To describe the epidemiology of CNS infections in Singapore.
2. To improve the diagnosis of aetiologies of CNS infections through a systematic clinical, laboratory and neuro-radiological evaluation and extensive diagnostic testing.
3. To evaluate the prognosis, long-term outcomes and socio-economic costs of CNS infections.
4. To establish an archive of biological tissues from patients with encephalitis and CNS infections that can be utilized for future testing for emerging novel pathogens or non-infectious aetiologies.

The study will recruit 400 patients over 2 years from 5 restructured hospitals in Singapore. As this is not a comparative study, sample size was not determined.

The study involves clinical and laboratory data collection. Data will also be collected on quality of life and for health economic analysis. The quality of data and its integrity will be periodically reviewed by the Principal Investigator and members of the study team. All samples stored will be de-identified and all data will be de-identified during analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical suspicion for Central Nervous system (CNS) infections, OR
2. Any two of the following,

   1. Fever or history of fever (≥ 38 °C) during the presenting illness
   2. Seizures of new onset
   3. Focal neurological deficits
   4. Cerebrospinal fluid white cell count pleocytosis (> 4 White blood cells (WBC)/uL)
   5. Abnormal neuroimaging suggestive of CNS infection.
   6. Abnormal electroencephalogram (EEG) suggestive of CNS infection
   7. Depressed or altered level of consciousness, OR
3. No alternative aetiology for acute paralysis identified (e.g stroke, trauma, myopathy etc)

Exclusion Criteria:

1. Patient or next of kin unwilling to give consent
2. Patients with indwelling ventricular devices such as EVD (external ventricular drain), VP (ventriculo-peritoneal) shunts

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient admitted to the hospital and who meets clinical case definition will be recruited in the study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of the various infective etiologies causing CNS infections in Singapore | 36 months
  Annual rates of the various infective causes from year 2013 to year 2016

SECONDARY OUTCOMES:
Clinical features of patients with CNS infections in Singapore | Between D1(day of recruitment)-D180(last day of follow up)
Clinical characteristics of patients diagnosed with CNS infections: . | Day1- Day180
  gender, presenting symptoms, duration between symptoms to diagnosis etc
Clinical course of patients with CNS infections, | Day1-Day180
  development of any complications and their long term outcomes/prognosis
Treatment modalities of the CNS infections | Day 1-Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Limin Wijaya, MD, Principal Investigator — SGH
Locations (1):
- Singapore General Hospital, Singapore, Singapore